CLINICAL TRIAL: NCT06438289
Title: Use of Ultrasound to Investigate Tip Dislodgment of Epicutaneous-caval Catheter: a Multicentric Study
Brief Title: Ultrasound to Investigate Tip Dislodgment of Epicutaneous-caval Catheter.
Acronym: DISLOTIP
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Francesco Raimondi, Professor, Federico II University
Other Study IDs: Protocol 335
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Migration of Implant or Internal Device
Keywords: tip location; ultrasound; epicutaneous-caval catheter; tip secondary migration; newborn; ECC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
This is a non-pharmacological, non-profit, prospective, observational multicenter study. Primarily, the study aims to demonstrate the feasibility of ultrasound methodology to study the secondary malposition of epicutaneous-caval catheters (ECC) in neonates.

After obtaining informed consent, the study involves performing ultrasound tip location on newborns who had an ECC placed. This will occur immediately after the placement and, if in a central position, subsequently at 60-120 minutes, 48-72 hours and 6-8 days post-placement. Data will be collected on various variables. Each Center will contribute at least 20 cases to the cohort and all data will be recorded in a database. The study is expected to last for 12 months

DETAILED DESCRIPTION:
Epicutaneous-caval catheters (ECCs) are among the most common central venous catheters used in neonatology. It is known that they can experience malpositioning over time from the moment of placement, leading to complications. In all studies conducted so far, tip location has been performed using X-ray. Ultrasound would be the ideal method for serial, bedside and radiatIon-free evaluation of ECC tip location to intercept any migrations. The primary endpoint of the study is to demonstrate the feasibility of ultrasound method for the assessment of secondary ECC malposition. Secondary endpoints include validating the results of previous Investigators monocentric study on the feasibility of ultrasound tip location applied to ECC and establishing the incidence of secondary malpositioning and the optimal timing for reassessing tip position after ECC placement. All neonates undergoing placement of 28 Gauge/1 French ECCs with a standardized securement system are included in the study, while neonates with major malformation are excluded. The study includes: obtaining written informed consent; performing ultrasound tip location using a standardized protocol (high right parasternal, apical four-chamber, short-axis left parasternal and bicaval subcostal views); If the tip is in a central position, repeating ultrasound tip location (using the same protocol) at 60-120 minutes, 48-72 hours and 6-8 days post-placement; collecting variables including sex, site of ECC insertion, weight at placement and at each tip location, postmenstrual age at placement and at each tip location, days of life at placement and at each tip location, respiratory support at placement and at each tip location, feasibility of ultrasound tip location for each ECC and for each specified time, ultrasound tip location result for each ECC and for each specified time and any displacement relative to the time of placement, as wall as any reported complications associated with secondary malpositioning. All ultrasound will be performed with the newborn in a standardized position: limb adducted and elbow extended if the catheter is placed from the upper limb, limb adducted and knee extended if the catheter is placed from the lower limb, neutral position if the catheter is placed from the scalp. The records of the ultrasound exams at each time for the first five cases enrolled by each Center will be sent to the Coordinator Center for evaluation of protocol compliance. Using the exact binomial method and setting a margin of error of 4% for a 95% of confidence interval, the investigators calculated that the sample size should be 196. The collected data will be recorded anonymously in an Excel database. Continuous variables will be expressed as means with minimum and maximum ranges, while categorical variables will be expressed as frequencies with percentages. Each case will be identified with an alphanumeric code to ensure data confidentiality. The principal investigator is the only person able to link the code to the identity of the patient. Parents, relative or guardians of eligible patients will be provided with all explanations regarding the experimental protocol by the study staff before enrollment. Information will be provided and parents will be given up to 12 hours to give their consent. The principal investigator will be responsible for the overall monitoring of data and the safety of the study participants. No funding or additional costs beyond common current practice are anticipated.

ELIGIBILITY:
Inclusion Criteria:

* neonates undergoing placement of 28 G/1 Fr ECCs with a standardized securement system

Exclusion Criteria:

* neonates with major malformation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: neonates undergoing placement of 28G/1 Fr ECCs with a standardized securement system
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of cases in which ultrasound tip location is feasible to study ECC secondary malposition | 8 days from the ECC placement
  percentage, from 0% to 100%

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Federico II- Neonatal Intensive Care Unit, Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Practice Guidelines for Central Venous Access 2020: An Updated Report by the American Society of Anesthesiologists Task Force on Central Venous Access. Anesthesiology. 2020 Jan;132(1):8-43. doi: 10.1097/ALN.0000000000002864. No abstract available. PMID 31821240
- [Background] Barone G, Pittiruti M. Epicutaneo-caval catheters in neonates: New insights and new suggestions from the recent literature. J Vasc Access. 2020 Nov;21(6):805-809. doi: 10.1177/1129729819891546. Epub 2019 Dec 5. PMID 31804149
- [Background] Costello JM, Clapper TC, Wypij D. Minimizing complications associated with percutaneous central venous catheter placement in children: recent advances. Pediatr Crit Care Med. 2013 Mar;14(3):273-83. doi: 10.1097/PCC.0b013e318272009b. PMID 23392365
- [Background] de Jonge RC, Polderman KH, Gemke RJ. Central venous catheter use in the pediatric patient: mechanical and infectious complications. Pediatr Crit Care Med. 2005 May;6(3):329-39. doi: 10.1097/01.PCC.0000161074.94315.0A. PMID 15857534
- [Background] Acun C, Baker A, Brown LS, Iglesia KA, Sisman J. Peripherally inserted central cathether migration in neonates: Incidence, timing and risk factors. J Neonatal Perinatal Med. 2021;14(3):411-417. doi: 10.3233/NPM-200684. PMID 33459671
- [Background] Gupta R, Drendel AL, Hoffmann RG, Quijano CV, Uhing MR. Migration of Central Venous Catheters in Neonates: A Radiographic Assessment. Am J Perinatol. 2016 May;33(6):600-4. doi: 10.1055/s-0035-1570341. Epub 2016 Jan 5. PMID 26731179
- [Background] Srinivasan HB, Tjin-A-Tam A, Galang R, Hecht A, Srinivasan G. Migration patterns of peripherally inserted central venous catheters at 24 hours postinsertion in neonates. Am J Perinatol. 2013 Nov;30(10):871-4. doi: 10.1055/s-0033-1333672. Epub 2013 Feb 4. PMID 23381907
- [Background] Grasso F, Capasso A, Pacella D, Borgia F, Salome S, Capasso L, Raimondi F. Ultrasound Guided Catheter Tip Location in Neonates: A Prospective Cohort Study. J Pediatr. 2022 May;244:86-91.e2. doi: 10.1016/j.jpeds.2021.12.059. Epub 2021 Dec 28. PMID 34971654
- [Derived] Grasso F, Capasso A, Dolce P, Ausanio G, Bernardo I, Poggi C, Dani C, Bonadies L, Baraldi E, Landi M, Tomasini B, Spagnuolo F, Carpentieri M, D'Andrea V, Vento G, Rodriguez-Perez C, Risso FM, Barone G, Ancora G, Ficial B, Biban P, Pittiruti M, Capasso L, Raimondi F. Ultrasound-guided tip location and detection of tip migration of neonatal peripherally inserted central catheters: a prospective, multicenter study (DISLOTIP study). Crit Care. 2025 Dec 20;29(1):532. doi: 10.1186/s13054-025-05800-1. PMID 41422244